CLINICAL TRIAL: NCT06732830
Title: Clinical Trial for the Evaluation of I+Med's DayDrop Advanced Ophthalmic Drop in Improving Signs and Symptoms of Mild/Moderate Dry Eye
Brief Title: Clinical Trial to Assess the Effectiveness of I+Med's DayDrop Advanced Ophthalmic Drop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i+Med S.Coop. (Industry)
Collaborators: Bioaraba Health Research Institute (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDROPA-PIC01-2021
Record Dates: First submitted 2024-03-05; First posted 2024-12-13 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Syndrome
Keywords: Dry eye; DayDrop; Ophtalmic Tears
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Quasi-experimental before-after clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DayDrop Advanced (Experimental): Participants will use DayDrop Advanced every day.
  Interventions: Device: DayDrop Advanced ophthalmic drop

INTERVENTIONS:
Device: DayDrop Advanced ophthalmic drop — The patient will administer 1 or 2 drops of DayDrop Advanced in each eye 3 times a day for 3 months.

SUMMARY:
Clinical trial conducted with the aim of evaluating changes in the signs of dry eye through the change in the amount of tears produced, measured through the Schirmer test. It will be performed in 45 patients diagnosed with mild/moderate dry eye who meet the inclusion/exclusion criteria. Follow-up will be 12 weeks with a maximum of 4 visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes over 18 years of age.
* Patients diagnosed with mild-moderate dry eye who meet the following characteristics: Schirmer test ≥3 and ≤ 10 mm; BUT test ≥5 and ≤ 10 seconds and OSDI ≥13 and ≤ 33.
* Patients without other ophthalmologic pathologies.
* Have ability to self-administer drops.
* Have ability to understand the Patient Information Sheet.
* Sign the Informed Consent.

Exclusion Criteria:

* Patients diagnosed with severe dry eye.
* Ingestion of parasympathomimetic or antipsychotic medications .
* Glaucoma.
* Previous cataract surgery.
* Systemic treatment with corticosteroids or topical treatment with any ophthalmic medication except artificial tears in the week prior to the start of study treatment.
* Ocular infection or clinically significant inflammation.
* Ocular surgery in the 3 months prior to the study.
* Sjögren's syndrome.
* Stevens-Johnson syndrome.
* History of allergic conjunctivitis.
* Pregnancy or planned lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Changes in the intensity of dry eye measured by Schirmer's test. | At baseline, in week 4 and in week 12
  The Schirmer test measures the amount of tears produced in mm of wetted strip.A greater distance in the Schirmer test implies a higher amount of tears produced and therefore a lower intensity of dry eye.

SECONDARY OUTCOMES:
Changes in dry eye signs through modifications in tear film thickness measured by Optical Coherence Tomography. | At baseline, in week 4 and in week 12
  Optical Coherence Tomography (OCT) evaluates changes in dry eye signs through changes in the thickness of the tear film, measured in microns.
Changes in dry eye signs through the tear breakup time measured by TBUT test. | At baseline, in week 4 and in week 12
  The TBUT test measures the tear break-up time (seconds until the appearance of tear break-up). Normal values are considered to be 10 seconds or more. The values from both eyes will be collected, and an average will be calculated for analysis.
Changes in dry eye symptoms through the OSDI scale. | At baseline, in week 4 and in week 12
  The OSDI scale allows for the assessment of the severity and classification of dry eye. The test results are classified as ≤13 normal, between 13 and 22 mild/moderate, and between 23 and 50 moderate/severe.
Satisfaction with Treatment. | At Week 12
  Pacient´s satisfaction with the treament as assessed using a brie survey. Possible responses range from not satisfied, indifferent, satisfied, very satisfied, and exceptionally satisfied.
Adverse events. | Through study completion, apprroximately 12 weeks
  Evaluating number and severity of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Araba, Vitoria-Gasteiz, Álava, Spain